CLINICAL TRIAL: NCT00422149
Title: Twin SUBLIVAC® Grasses Clinical Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: H.A.J. Kleinjans, HAL Allergy BV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG/0021; EudraCTnr: 2005-005175-16
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic
Keywords: Sublingual immunotherapy; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): SUBLIVAC® Grasses treatment
  Interventions: Drug: SUBLIVAC® Grasses/Placebo treatment; Drug: SUBLIVAC® Grasses treatment
- 2 (Placebo Comparator): Placebo treatment
  Interventions: Drug: SUBLIVAC® Grasses/Placebo treatment; Drug: Placebo treatment

INTERVENTIONS:
Drug: SUBLIVAC® Grasses/Placebo treatment — SUBLIVAC® Grasses/Placebo treatment
Drug: SUBLIVAC® Grasses treatment — SUBLIVAC® Grasses treatment
  Arms: 1
Drug: Placebo treatment — Placebo treatment
  Arms: 2

SUMMARY:
To show that treatment with SUBLIVAC® Grasses is clinically effective by means of reduction in allergic symptoms and/or use of allergic symptomatic medication in subjects suffering from IgE mediated allergic complaints triggered by grass pollen.

DETAILED DESCRIPTION:
Indication under study: IgE mediated allergic disorders triggered by grass pollen.

Number of centres: approximately 50.

Study period planned: Q2-2006 until Q3-2008 Analysis after one exposed season (2007); based on the outcome the study will be stopped or continued for another season.

Subject selection criteria: Seasonal rhinitis and/or rhinoconjunctivitis with or without mild asthma (FEV1 > 70%) related to grass pollen, age 12 years or older.

Dosage schedule: Start with two drops daily of SUBLIVAC® and increase by two drops daily, until the maintenance dose of 10 drops SUBLIVAC® GrassesSUBLIVAC® Grasses is reached.

Route of administration: Sublingual application (drops are to be held underneath the tongue for 2-3 minutes and then will be swallowed).

Duration of treatment: 6 to 12 months blinded per subject . Efficacy parameters

ELIGIBILITY:
Inclusion Criteria:

* Subjects with allergic rhinoconjunctivitis with or without mild asthma FEV1 ≥ 70%) for at least 2 years. Their allergic symptoms should be related to grass pollen Use of anti-allergy symptomatic medication in the last pollen season (or, in case of a low pollen season, in one of the two previous years)
* A positive skin prick test (>3 mm) for early flowering treesgrasses and specific serum IgE-test(>1 U/ml) for grass pollen (Lolium perenne, Phleum pratense and Poa pratensis).

Exclusion Criteria:

* A positive SPT for perennial allergens of house dust mite
* Allergy to any of the excipients
* Symptoms related to concomitant sensitisation to perennial allergens of pets
* Chronic asthma or emphysema, particularly with a FEV1 < 70 % of predicted value or use of inhalation corticosteroids outside grass and tree pollen season for more than two episodes and/or longer than fourteen days
* Use of symptomatic medication for more than three episodes and/or longer than three days outside the tree- or grass pollen season
* Serious immuno-pathological diseases or malignancies (including auto-immune diseases, tuberculosis, HIV)
* Inflammation and infection of the target organ
* Severe atopic dermatitis requiring systemic immuno-suppressive medication
* Allergen specific immuno-therapy treatment within the last 5 years for a period longer than three months
* History of life threatening anaphylactic events, including anaphylactic food allergy, insect venom anaphylaxis, exercise or drug induced anaphylaxis
* A positive pregnancy test, lactation or inadequate contraceptive measures Alcohol- or drug abuse
* Lack of co-operation or severe psychological disorders

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical index score (CIS), measured during the pollen season, in the treatment group compared to the placebo group. | June, July, August 2007

SECONDARY OUTCOMES:
CIS derived variables | June, July and August 2007
RQLQ, quantitative skin prick test | Pollen season 2006 and 2007
oral allergy syndrome | October 2006 until September 2007
mast-cell serum tryptase | 6 months therapy
specific immunoglobulins (IgE and IgG). | 6 months therapy

CONTACTS AND LOCATIONS:
Overall Officials: R Peter, Prof.Dr.med, Principal Investigator — Zentrum für Klinische Forschung, Helholzstrasse 8/1, 89081 Ulm, Germany
Locations (59):
- Belgium (7):
  - Dr. P. van Durme, Antwerp
  - Centrum Gespecialiseerde Geneeskunde Genk, Genk
  - UZ Gent, Dienst NKO, 1P1, Ghent
  - UZ Gasthuisberg, Afd. Allergie/Immunologie, Leuven
  - UZ Gasthuisberg, Dienst Kindergeneeskunde, Leuven
  - UZ Gasthuisberg, lokatie St. Rafaël, Leuven
  - Kinderallergie-Astma kinderz., Mechelen
- Germany (27):
  - Allergologie Aachen, Aachen
  - Charité - Universitätsmedizin Berlin, Berlin
  - Studienzentrum Berlin, Berlin
  - Allergologie Braunschweig, Braunschweig
  - Priv.-Doz. Hals-Nasen-Ohrenheilkunde plastische Operationen Allergologie, Darmstadt
  - Allergologie Dorsten, Dorsten
  - Hals, Nasen- u. Ohrenheilkunde Dortmund, Dortmund
  - Hals, Nasen- u. Ohrenheilkunde Duisburg, Duisburg
  - Medi-Center Düren, Düren
  - Hals, Nasen- u. Ohrenheilkunde Düsseldorf, Düsseldorf
  - Heinrich-Heine-Universität Düsseldorf, Hautklinik, Düsseldorf
  - Universität Erlangen, Poliklinik für Kinder und Jugendliche, Erlangen
  - Gemeinschaftspraxis Dr. M. Feldmann und Dr. N. Karadiakos, Essen
  - Hals, Nasen- u. Ohrenheilkunde Essen, Essen
  - Allergologie Gifhorn, Gifhorn-Winkel
  - Drobnitzky Franz-Josef Dr.med. Kinderarzt-Allergologie und Frank-Peter Dr.med. Kinderarzt-Neonatologie Gemeinschaftspraxis, Gütersloh
  - Klinik für Pneumologie, Intensiv- und Schlafmedizin Klinikum, Hanover
  - Med.Hochschule Hannover, Kinderklinik, Hanover
  - Allergologie Jülich, Jülich
  - Allergologie Kassel, Kassel
  - HNO - Krefeld, Krefeld
  - Hals, Nasen- u. Ohrenheilkunde Lüdenscheid, Lüdenscheid
  - Allgemeinmedizin Stockach, Baden, Stockach
  - Zentrum für Klinische Forschung, Helmholtzstrasse 8/1, 89081 Ulm, Germany, Ulm
  - Gemeinschaftspraxis für HNO Heilkunde, Allergologie und plastische Chirurgie, Wiesbaden
  - Hals, Nasen- u. Ohrenheilkunde Willich, Willich
  - Gemeinschaftspraxis für Hals-Nasen-Ohrenheilkunde, Wuppertal
- Netherlands (4):
  - Meander Medisch Centrum, lokatie Baarn, Afdeling KNO, Amersfoort
  - Allergologen Maatschap Arnhem, Arnhem
  - Wilhelmina Ziekenhuis Assen, Afdeling KNO, Assen
  - Vlietland Ziekenhuis, lokatie Schiedam, KNO, Schiedam
- Poland (21):
  - Medical University of Bialystok, Department of Pediatrics and Allergology, Bialystok
  - Medical University of Gdansk, Department of Allergology, Gdansk
  - FARMA-MED. Sp. z o. o., Inowrocław
  - Jagiellonian University Medical College, Department of Allergy and Immunology, Krakow
  - Jagiellonian University Medical College, Department of Allergology and Dermatology, Krakow
  - Klinika Pneumonologii i Alergologii Uniwersytet Medyczny w Lodzi, Lodz
  - NZOZ Centrum Alergologii, Lodz
  - Medical University of Lodz, Department of Allergology and Pulmonology, Lodz
  - Medical University of Lodz, Department of Clinical Immunology and Allergy, Lodz
  - Medical University of Lodz, Department of Pediatrics and Allergology, Lodz
  - Medical University of Lublin, Department of Allergology and Immunotherapy, Lublin
  - Klinika Pneumonologii Onkologii i Alergologii SPSK Nr 4, Lublin
  - Oddzial Dzieciecy SPZOZ, Pabianice
  - Institute of Allergy and Lung Disease Rabka, Department of Allergology and Pneumonology, Rabka-Zdrój
  - Specjalistyczny Zespól Diagnostyczno-Konsultacyjny Problemów Alergii Emil Florkiewicz, Sieradz
  - Gabinet Lekarski Bozena Kubicka-Kozik Poradnia Alergologiczna, Tomaszów Mazowiecki
  - Specjalistyczny Niepubliczny Zaklad Leczenia Alergii i Diagnostyki Alergologicznej IRMED 2, Warsaw
  - Military Institute of the Health Services, Department of Infection Disease and Allergology, Warsaw
  - Military Institute of the Health Services, Department of Internal Disease Pulmonology and Allergology, Warsaw
  - Medical University of Wroclaw, Department of Internal Disease and Allergology, Wroclaw
  - Medical University of Silesia, Department of Internal Disease, Allergology and Clinical Immunology, Zabrze